CLINICAL TRIAL: NCT01927575
Title: Pilot Study Comparing Diagnostic Imagining Versus FujiFilm's Digital Radiographic AcSellerate CsI System With Tomosynthesis
Brief Title: Pilot Study Comparing Diagnostic Imaging Versus Tomosynthesis in Detection of Hip, Wrist or Tibia Injury
Acronym: TOMO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to close trial
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FMSU2012-001
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Wrist Injury; Tibial Fracture; Hip Injury
Keywords: TOMOSYNTHESIS
MeSH Terms: conditions — Wrist Injuries; Tibial Fractures; Hip Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard X-Ray + CT (Active Comparator): Standard X-Ray + CT arm to be used as comparative arm for investigational imaging device. Investigators will determine standard of care to be used on a per subject basis.
  Interventions: Device: Standard X-Ray + CT; Device: TOMO
- Standard X-Ray + MRI (Active Comparator): Standard X-Ray + MRI arm to be used as comparative arm for investigational imaging device. Investigators will determine standard of care to be used on a per subject basis.
  Interventions: Device: Standard X-Ray + MRI; Device: TOMO
- Tomo (Experimental): Fujifilm Digital Radiographic AcSelerate CsI System with Tomosynthesis
  Interventions: Device: Standard X-Ray + CT; Device: Standard X-Ray + MRI; Device: TOMO

INTERVENTIONS:
Device: Standard X-Ray + CT — Standard of Care X-Ray Imaging + CT
  Arms: Standard X-Ray + CT; Tomo
Device: Standard X-Ray + MRI — Standard of Care X-Ray Imaging + MRI
  Arms: Standard X-Ray + MRI; Tomo
Device: TOMO — Fujifilm Digital Radiographic AcSelerate CsI System with Tomosynthesis

SUMMARY:
To acquire and build a library of image sets to determine if Fuji's TOMO imaging device can replace or compliment current imaging standards to assess patients with hip, wrist or tibia injuries.

DETAILED DESCRIPTION:
Subjects presenting with a wrist injury, tibial fracture, or hip injury that require protocol defined standard imaging will have an X-Ray, CT Scan (or MRI per site preference) and TOMO completed. Images will be assessed to determine if TOMO is appropriate to supplement or replace the need for the other standard images.

ELIGIBILITY:
Inclusion Criteria:

* Physician request to have diagnostic imaging for condition areas

Exclusion Criteria:

* Under 18
* Pregnancy
* Insufficient Anatomical Coverage or Potential Image Problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Bova, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University of Chicago, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who present for, are undergoing, or have undergone 'standard of care' general x-ray and CT or MRI examinations, which meet all of the study enrollment criteria, may be approached and enrolled. Each subject would then have a 3rd image taken using Fujifilm's Digital Radiographic AcSelerate CsI System with Tomosynthesis.
Pre-assignment Details: Subjects are recruited as long as they had either an x-ray and CT or an x-ray and MRI, and sign a consent to have a third image taken with Fujifilm's Digital Radiographic AcSelerate CsI System with Tomosynthesis.
Groups:
- All Study Participants: Standard of care X-Ray imaging plus CT to be compared with research imaging device.
  Standard X-Ray: Standard of Care X-Ray Imaging + CT
  Followed by Tomo Imaging
Period: Overall Study
Arm/Group | All Study Participants
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 patient was enrolled in this study, and they underwent Standard X-Ray and CT as well as Tomosynthesis.
Groups:
- All Study Participants: Standard X-Ray + CT arm to be used as comparative arm for investigational imaging device. Investigators will determine standard of care to be used on a per subject basis.
  Standard X-Ray + CT: Standard of Care X-Ray Imaging + CT
  Followed by Tomo Imaging
Arm/Group | All Study Participants
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (NA) — No SD able to be calculated due to only 1 patient enrolled.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Whom Tibia Injury Was Detected
Description: Clinical utility where the DTS could replace and/or complement existing imaging procedures; for example, Computed Tomography for fractures of the tibial plateau or scaphoid - where radiation dose, access to modality and cost play a factor in planning initial diagnosis and/or follow-up imaging strategies. Subsequent independent review by the principal investigator (PI) [or designee] to show the ability of the Fujifilm DTS system to provide images of clinical equivalence compared to those acquired on other FDA cleared imaging systems.
Time Frame: Baseline Imaging Collection
Population: Three sets (1 - X-ray, 1- CT and 1 - Digital Tomosynthesis) of images of the tibia evaluated to confirm acceptable image quality and provided clinical and diagnostic value.
Measure: Number; unit: participants
Groups:
- Standard X-Ray: Standard of care X-Ray imaging to be compared with research imaging device.
  Followed by Tomo imaging
  No AE's
- Standard CT: Standard of care CT imaging to be compared with research imaging device.
  Followed by Tomo imaging
  No AE's
- Tomosynthesis: Tomosynthesis imaging to be compared to standard of care CT and X-ray
  No AEs
Arm/Group | Standard X-Ray | Standard CT | Tomosynthesis
Number analyzed (Participants) | 1 | 1 | 1
participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 day; Standard of Care X-ray, CT and Tomo all completed within this day.
Groups:
- Standard X-Ray; Standard CT; Tomo: Standard of care X-Ray, and CT imaging to be compared with research imaging device.
  Standard X-Ray: Standard of Care X-Ray Imaging
  Followed by Tomo imaging
Arm/Group | Standard X-Ray | Standard CT | Tomo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No